CLINICAL TRIAL: NCT04364867
Title: Randomized Clinical Trial of Exparel vs Pain Pump for Post-operative Pain Control After Total Shoulder Arthroplasty
Brief Title: Exparel for Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norton Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-N0122
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2022-06

CONDITIONS: Total Shoulder Arthroplasty
Keywords: Total Shoulder Arthroplasty; Post-operative Pain; Pain pump; Liposomal Bupivacaine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Experimental): Single shot Exparel 10cc (133mg) mixed with 10cc of 0.5% Bupivicaine
  Interventions: Drug: Exparel
- Pain pump (Active Comparator): Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the Post Anesthesia Care Unit infusing at 4cc/hr. The patient will go home with that device until it runs out.
  Interventions: Drug: Pain Pump

INTERVENTIONS:
Drug: Exparel — Single shot Exparel 10cc (133mg) mixed with 10cc of 0.5% Bupivicaine
  Arms: Exparel
Drug: Pain Pump — Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the Post Anesthesia Care Unit infusing at 4cc/hr. The patient will go home with that device until it runs out.
  Arms: Pain pump

SUMMARY:
The primary objective of this study is to determine if Exparel leads to better pain scores at 24, 48 and 72 hours after Total Shoulder Arthroplasty (TSA) compared to a pain pump. Secondary objectives are (1) to determine if patients on Exparel use less narcotics and (2) have earlier return of functional use of the involved arm after surgery compared to the pain pump and (3) if use of Exparel leads to cost savings

METHODS

Sample size:

Based on prior studies on anesthetics for TSA, the mean worst pain score in the 24 hours after surgery was 5.4, based on a 0 to 10 scale. To detect a change of 2 points, alpha of 0.05, beta of 0.80, a sample size of 51 subjects in each group will be required. To account for drop-outs, a total of 60 subjects in each arm will be enrolled.

Inclusion criteria Patients undergoing unilateral primary TSA or reverse TSA Indication for surgery is osteoarthritis, rotator cuff arthropathy or massive irreparable rotator cuff tears Surgery performed by the Principal Investigator Anesthesia administered by Co-Principal Investigator Willing and able to sign an Informed Consent Exclusion criteria Indication for surgery is fracture Comorbid psychiatric diagnosis requiring therapy and/or medication except anxiety or depression Comorbid chronic pain syndrome (reflex sympathetic dystrophy, fibromyalgia) Has hepatic disease On workers compensation/disability/litigation Known adverse reaction to medications to be administered On long-acting narcotic pain medication (including extended release narcotic pain medications and methadone) Home Oxygen requirement whether as needed or scheduled. Contralateral Phrenic Nerve paralysis / incompetence. Body Mass Index ≥ 50 Randomization will be a varied blocked randomization with blocks of 12, 15 and 18 using sealed envelopes

Treatment arms:

Control: Pain catheter based pain control. Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the Post Anesthesia Care Unit infusing at 4cc/hr. The patient will go home with that device until it runs out.

Interventional: Single shot Exparel 10cc (133mg) mixed with 10cc of 0.5% Bupivicaine

Both arms will receive the same multimodal analgesia medications preoperatively. Celebrex 400mg PO, Gabapentin 600mg PO, Tylenol 1 gram PO, unless contraindicated.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if Exparel leads to better pain scores at 24, 48 and 73 hours after TSA compared to a pain pump. Secondary objectives are (1) to determine if patients on Exparel use less narcotics and (2) have earlier return of functional use of the involved arm after surgery compared to the pain pump and (3) if use of Exparel leads to cost savings

METHODS

Sample size:

Based on prior studies on anesthetics for TSA, the mean worst pain score in the 24 hours after surgery was 5.4, based on a 0 to 10 scale. To detect a change of 2 points, alpha of 0.05, beta of 0.80, a sample size of 51 subjects in each group will be required. To account for drop-outs, a total of 60 subjects in each arm will be enrolled.

Inclusion criteria Patients undergoing unilateral primary TSA or reverse TSA Indication for surgery is osteoarthritis, rotator cuff arthropathy or massive irreparable rotator cuff tears Surgery performed by the Principal Investigator Anesthesia administered by Co-Principal Investigator Willing and able to sign an Informed Consent Exclusion criteria Indication for surgery is fracture Comorbid psychiatric diagnosis requiring therapy and/or medication except anxiety or depression Comorbid chronic pain syndrome (reflex sympathetic dystrophy, fibromyalgia) Has hepatic disease On workers compensation/disability/litigation Known adverse reaction to medications to be administered On long-acting narcotic pain medication (including extended release narcotic pain medications and methadone) Home Oxygen requirement whether as needed or scheduled. Contralateral Phrenic Nerve paralysis / incompetence. Body Mass Index ≥ 50 Randomization will be a varied blocked randomization with blocks of 12, 15 and 18 using sealed envelopes

Treatment arms:

Control: Pain catheter based pain control. Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the Post Anesthesia Care Unit infusing at 4cc/hr. The patient will go home with that device until it runs out.

Interventional: Single shot Exparel 10cc (133mg) mixed with 10cc of 0.5% Bupivicaine

Both arms will receive the same multimodal analgesia medications preoperatively. Celebrex 400mg PO, Gabapentin 600mg PO, Tylenol 1 gram PO, unless contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TSA or reverse TSA
* Indication for surgery is osteoarthritis, rotator cuff arthropathy or massive irreparable rotator cuff tears
* Surgery performed by the Principal Investigator
* Anesthesia administered by Co-Principal Investigator
* Willing and able to sign an Informed Consent

Exclusion criteria

* Indication for surgery is fracture
* Comorbid psychiatric diagnosis requiring therapy and/or medication except anxiety or depression
* Comorbid chronic pain syndrome (reflex sympathetic dystrophy, fibromyalgia)
* Has hepatic disease
* On workers compensation/disability/litigation
* Known adverse reaction to medications to be administered
* On long-acting narcotic pain medication (including extended release narcotic pain medications and methadone)
* Home Oxygen requirement whether as needed or scheduled.
* Contralateral Phrenic Nerve paralysis / incompetence.
* Body Mass Index ≥ 50

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Krupp, MD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Healthcare, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Pump: Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the PACU infusing at 4cc/hr. The patient will go home with that device until it runs out.
  Pain Pump: Subject will receive an interscalene block with Ropivicaine 0.5% (20cc), and then a pain pump attached in the PACU infusing at 4cc/hr. The patient will go home with that device until it runs out.
Period: Overall Study
Arm/Group | Exparel | Pain Pump
Started | 51 | 51
Completed | 19 | 35
Not Completed | 32 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Pain Pump | Total
Number analyzed (Participants) | 19 | 35 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (6.96) | 67.15 (7.17) | 66.68 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 25
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 18 | 33 | 51
  Race: African American | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 35 | 54

OUTCOME MEASURES:

1. Primary Outcome: Pain Score in the 24 Hours After Surgery
Description: Worst pain score (0 [none] to 10 [worst possible]) in the 24 hours after surgery
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
score on a scale | 0.76 (0.97) | 3.37 (2.86)

2. Secondary Outcome: Pain Score in the 48 Hours After Surgery
Description: Worst pain score (0 [none] to 10 [worst possible]) in the 48 hours after surgery
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
score on a scale | 2.53 (1.42) | 4.70 (3.23)

3. Secondary Outcome: Cumulative Morphine Milligram Equivalents at 24 Hours
Description: Cumulative Morphine Milligram Equivalents consumed at 24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
Morphine Milligram Equivalents (MME) | 4.58 (6.53) | 3.57 (3.84)

4. Secondary Outcome: Cumulative Morphine Milligram Equivalents at 48 Hours
Description: Cumulative Morphine Milligram Equivalents consumed at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
Morphine Milligram Equivalents (MME) | 4.58 (0.88) | 4.19 (0.72)

5. Secondary Outcome: Cumulative Morphine Milligram Equivalents at 72 Hours
Description: Cumulative Morphine Milligram Equivalents consumed at 72 hours
Time Frame: 72hours
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
Morphine Milligram Equivalents (MME) | 4.58 (00.88) | 4.31 (0.65)

6. Secondary Outcome: Pain Score in the 72 Hours After Surgery
Description: Worst pain score (0 [none] to 10 [worst possible]) in the 72 hours after surgery
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exparel | Pain Pump
Number analyzed (Participants) | 19 | 35
score on a scale | 2.94 (2.73) | 3.69 (2.93)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Dislodgment of pain pump catheter
Arm/Group | Exparel | Pain Pump
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/35
Other Adverse Events (participants affected / at risk) | 0/19 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel (N=19) | Pain Pump (N=35)
Catheter Dislodgement (Product Issues) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT04364867/Prot_SAP_001.pdf